CLINICAL TRIAL: NCT01089439
Title: Nitric Oxide Therapy for Acute Chest Syndrome in Sickle Cell Disease Children: Randomized, Double Blind Placebo-controlled Concept-proof Trial
Brief Title: Nitric Oxide Therapy for Acute Chest Syndrome in Sickle Cell Disease Children
Acronym: INNOSTAPED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P071003
Record Dates: First submitted 2009-10-21; First posted 2010-03-18 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2013-08

CONDITIONS: Acute Chest Syndrome; Sickle Cell Disease
Keywords: Nitric oxide
MeSH Terms: conditions — Acute Chest Syndrome; Anemia, Sickle Cell | interventions — Endothelium-Dependent Relaxing Factors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1: INOMAX (Active Comparator): Nitric oxide by inhalation INOMAX:
  active arm treated with nitric oxide
  Interventions: Drug: Nitric oxide by inhalation INOMAX
- 2: Placebo (Placebo Comparator): placebo arm treated with placebo at the same conditions
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitric oxide by inhalation INOMAX — Nitric oxide by inhalation INOMAX 800 ppm
  40 ppm during 24 hours then 20 ppm during 24 hours then 10 ppm during 24 hours
  Other Names: INOMAX
  Arms: 1: INOMAX
Drug: Placebo — placebo
  Arms: 2: Placebo

SUMMARY:
Acute chest syndrome is a severe sickle cell disease complication in children requiring blood transfusion therapy to prevent acute respiratory failure and death. Nitric oxide is a potent vasodilator that could reverse pulmonary vascular occlusion and restore normal oxygenation. The randomized trial will test that hypothesis.

DETAILED DESCRIPTION:
Acute chest syndrome is a severe sickle cell disease complication in children requiring blood transfusion therapy to prevent acute respiratory failure and death. Nitric oxide is a potent vasodilator that could reverse pulmonary vascular occlusion and restore normal oxygenation. The randomized trial will test that hypothesis in a prospective randomized double-blind placebo controlled study. 50 children in two years will be included: 25 in each arm.

ELIGIBILITY:
Inclusion Criteria:

* child between 1 and 18 years old
* Sickle cell anemia or equivalent (sickle beta 0 thalassemia)whoe weight is between 10kg and 65kg
* presenting acute chest syndrome as defined a new radiological infiltrate with tachypnea, respiratory discomfort, cough, chest wall pain and fever more than 38.5°C
* hypoxaemia with transcutaneous oxygen saturation equal or less than 92%
* informed consent signed by parents and approved by the child able to express his consent
* insured by the National social security system or by the universal medical insurance
* previous medical physical examination

Exclusion Criteria:

* respiratory distress with hypoxaemia with transcutaneous oxygen saturation equal or less than 92% under more than 5l/min of oxygen or 40% oxygen inhaled, hypercapnia signs 'sweating, altered consciousness, paCO2 more than 60mmHg) with need of emergency exchange transfusion and/or tracheal intubation with mechanical ventilation
* Isolated acute asthmatic crisis
* stroke or priapism with emergency acute transfusion needed
* acute anemia with hemoglobin drop of more than 20% as compared to steady state hemoglobin
* chronic long term transfusion therapy
* nitric oxyde hypersensitivity
* patients with right-left extra-pulmonary cardiac shunt
* patient previously included in the protocol
* patient participating in another interventional protocol
* pregnancy or breast feeding

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2010-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
We will observe the patient's transfusional needs under nitric oxide (MONOXYDE AZOTE) versus placebo inhaled therapy to evaluate inhaled MOXYDE AZOTE efficacy on improving oxygenation (transcutaneous O2 superior to 92% ) | Oxygenation improvement (transcutaneous O2 superior to 92%) after Gas inhalation will be evaluate 2hours after inclusion and therafter every 2 hours until 12 hours therapy and then every six hours for 3days and then once a day till hospital discharge

SECONDARY OUTCOMES:
Number of blood transfusions and total transfused blood volume | 7 to 10 days
Quantity of Pain-killer drugs required and particularly OPIOIDS | 7 to 10 days
Duration of Nitric oxide therapy | after 7 to 10 days
Duration of OXYGENOTHERAPY | 7 to 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Malika Benkerrou, Dr., Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hoipital Robert Debre, Paris, France